CLINICAL TRIAL: NCT02654080
Title: A Phase 1 Trial to Evaluate the Safety, Tolerability, and Immunogenicity of a Prime-Boost Regimen of HIV-1 Nef/Tat/Vif, Env pDNA Vaccine Delivered Intramuscularly With Electroporation and HIV-1 rVSV envC Vaccine in Healthy HIV-Uninfected Adult Participants
Brief Title: Evaluating the Safety, Tolerability, and Immunogenicity of a Prime-Boost Regimen of HIV-1 Nef/Tat/Vif, Env pDNA Vaccine Delivered Intramuscularly With Electroporation and HIV-1 rVSV envC Vaccine in Healthy, HIV-Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 112; 11988 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Genes, env

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Vaccine (Experimental): Participants will receive the HIV-1 nef/tat/vif, env pDNA vaccine at Day 0 and Months 1 and 3. They will receive the rVSV HIV envC vaccine boost at Months 6 and 9.
  Interventions: Biological: HIV-1 nef/tat/vif, env pDNA vaccine; Biological: rVSV HIV envC vaccine
- Group 2: Placebo (Placebo Comparator): Participants will receive placebo vaccine at Day 0 and Months 1, 3, 6, and 9.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: HIV-1 nef/tat/vif, env pDNA vaccine — 1500 mcg to be administered as 0.5 mL intramuscular (IM) in the deltoid of the non-dominant arm (unless medically contraindicated) using the Ichor Medical Systems TDS EP device
  Other Names: ProfectusVax DNA Plasmid HIV-1 nef/tat/vif, env
  Arms: Group 1: Vaccine
Biological: rVSV HIV envC vaccine — 1 × 10^7 PFU to be administered as 1 mL IM in the deltoid of the non-dominant arm (unless medically contraindicated)
  Other Names: ProfectusVaxVSV IN HIV envC
  Arms: Group 1: Vaccine
Biological: Placebo — Sodium Chloride for Injection, USP 0.9%;
  At Months 0, 1, and 3: administered as 0.5 mL IM in the deltoid of the non-dominant arm (unless medically contraindicated) using the Ichor Medical Systems TDS EP device.
  At Months 6 and 9: administered as 1 mL IM in the deltoid of the non-dominant arm (unless medically contraindicated).
  Arms: Group 2: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of an HIV-1 nef/tat/vif, env pDNA vaccine delivered with electroporation (EP), followed by a recombinant vesicular stomatitis virus (rVSV) HIV envC vaccine boost, in healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
This study will evaluate the safety and tolerability of an HIV-1 nef/tat/vif, env pDNA vaccine delivered with EP, followed by a rVSV HIV envC vaccine boost, in healthy, HIV-uninfected adults.

Participants will be randomly assigned to one of two groups. Participants in Group 1 will receive the HIV-1 nef/tat/vif, env pDNA vaccine at Day 0 and Months 1 and 3, followed by the rVSV HIV envC vaccine boost at Months 6 and 9. Participants in Group 2 will receive placebo vaccine at Day 0 and Months 1, 3, 6, and 9. Study visits will occur at Day 0, Week 2, and Months 1, 1.5, 3, 3.25, 3.5, 6, 6.25, 6.5, 9, 9.25, 9.5, 12, and 15. Visits may include physical examinations, urine collection, blood collection, HIV testing, risk reduction counseling, assessments, and questionnaires. Participants will be contacted by study staff for follow-up monitoring annually for 3 years following the initial study injection.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria:

* Age of 18 to 50 years
* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Willing to be contacted annually after completion of scheduled clinic visits for a total of 3 years following initial study injection
* Agrees not to enroll in another study of an investigational research agent prior to completion of last required protocol clinic visit (excludes annual health contacts for safety surveillance)
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit

Laboratory Inclusion Values:

Hemogram/Complete Blood Count (CBC):

* Hemoglobin greater than or equal to 11.0 g/dL for volunteers who were born female, greater than or equal to 13.0 g/dL for volunteers who were born male
* White blood cell count equal to 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3

Chemistry:

* Chemistry panel: ALT, AST, and alkaline phosphatase less than 1.25 times the institutional upper limit of normal; creatinine less than or equal to institutional upper limit of normal; CPK less than or equal to 2.0 times the institutional upper limit of normal

Virology:

* Negative HIV-1 and -2 blood test: U.S. volunteers must have a negative FDA-approved enzyme immunoassay (EIA)
* Negative hepatitis B surface antigen (HBsAg)
* Negative anti-hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine:

* Normal urine:

  * Negative urine glucose, and
  * Negative or trace urine protein, and
  * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range)

Reproductive Status:

* Volunteers who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* Reproductive status: A volunteer who was born female must:

  * Agree to consistently use effective contraception (see protocol for more information) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception is defined as using the following methods:
  * Condoms (male or female) with or without a spermicide,
  * Diaphragm or cervical cap with spermicide,
  * Intrauterine device (IUD),
  * Hormonal contraception,
  * Any other contraceptive method approved by the HVTN 112 Protocol Safety Review Team (PSRT), or
  * Successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
  * Or be sexually abstinent.
* Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

General:

* Allergy to amide-type local anesthetics (bupivacaine [Marcaine], lidocaine [Xylocaine], mepivacaine [Polocaine/Carbocaine], etidocaine [Duranest], prilocaine [Citanest, EMLA® cream])
* Presence of implanted electronic medical device (e.g., pacemaker, implantable cardioverter defibrillator)
* Presence of surgical or traumatic metal implant in the upper limb and/or upper torso
* Sinus bradycardia (defined as less than 50 bpm on exam) or a history of cardiac arrhythmia: e.g., supraventricular tachycardia, atrial fibrillation, or frequent ectopy
* Neurological or neuropsychiatric disorder that may interfere with the assessment of safety: e.g., frequent recurring headaches (i.e., a pattern of greater than 1 headache per month affecting activities of daily living (ADLs)/work, frequent or severe/complicated migraines, cluster headaches), a chronic pain syndrome, dizziness, history of meningitis or encephalitis, cranial/spinal/peripheral neuropathy, limb weakness or paralysis, movement disorder, narcolepsy, stroke with sequelae, moderate/severe major depressive disorder, moderate/severe bipolar disorder
* Deltoid skin fold measurement by caliper greater than 40 mm
* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) greater than or equal to 40; or BMI greater than or equal to 35 with 2 or more of the following: age greater than 45, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, known hyperlipidemia
* Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing during the planned duration of the HVTN 112 study
* Pregnant or breastfeeding
* Active duty and reserve U.S. military personnel

Vaccines and Other Injections:

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 112 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 112 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 112 PSRT on a case-by-case basis.
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 28 days after injection (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (e.g., tetanus, pneumococcal, hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination

Immune System:

* Immunosuppressive medications received within 168 days before first vaccination. (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses less than 2 mg/kg/day and length of therapy less than 11 days with completion at least 30 days prior to enrollment.)
* Serious adverse reactions to vaccines or to vaccine components, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 90 days before first vaccination
* Autoimmune disease
* Immunodeficiency

Clinically Significant Medical Conditions:

* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report).

  * Exclude a volunteer who:
  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses moderate/high dose inhaled corticosteroids, or
  * In the past year has either of the following:
  * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
  * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these volunteers, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure. or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-03; Primary Completion 2017-08-24 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Frequency of local injection/EP site and systemic reactogenicity signs and symptoms | Measured through Month 15
Severity of local injection/EP site and systemic reactogenicity signs and symptoms | Measured through Month 15
Frequency of adverse events (AEs) | Measured through Month 15
  Categorized by MedDRA body system, MedDRA preferred term, severity and assessed relationship to study products. Detailed description of all AEs meeting Division of AIDS (DAIDS) criteria for expedited reporting.
Composite of safety laboratory measures: white blood cells (WBCs), neutrophils, lymphocytes, hemoglobin, alkaline phosphatase, platelets, alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine, and creatine phosphokinase (CPK) | Measured through Month 15
Magnitude of local injection/EP site pain as measured by a visual analog scale (VAS) | Measured through Month 15
Number of participants with early discontinuation of vaccinations and reasons for discontinuation | Measured through Month 15

SECONDARY OUTCOMES:
HIV-specific CD4+ T-cell response rates and magnitude 2 weeks after the last priming vaccination and 2 weeks after each boost | Measured through Month 9.5
HIV-specific CD8+ T-cell response rates and magnitude 2 weeks after the last priming vaccination and 2 weeks after each boost | Measured through Month 9.5
Magnitude and breadth of HIV-specific binding antibody responses as assessed by multiplex assay 2 weeks after each boost | Measured through Month 9.5
Neutralizing antibody magnitude and breadth against tier 1 and, if applicable, tier 2 HIV-1 isolates as assessed by area under the magnitude-breadth curves 2 weeks after each boost | Measured through Month 9.5

CONTACTS AND LOCATIONS:
Overall Officials: Greg Wilson, Study Chair — Vanderbilt University
Locations (2):
- United States (2):
  - Case Clinical Research Site, Cleveland, Ohio
  - Penn Prevention CRS, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Wilson GJ, Rodriguez B, Li SS, Allen M, Frank I, Rudnicki E, Trahey M, Kalams S, Hannaman D, Clarke DK, Xu R, Egan M, Eldridge J, Pensiero M, Latham T, Ferrari G, Montefiori DC, Tomaras GD, De Rosa SC, Jacobson JM, Miner MD, Elizaga M; HIV Vaccine Trials Network 112 Protocol Team. Cellular and humoral responses to an HIV DNA prime by electroporation boosted with recombinant vesicular stomatitis virus expressing HIV subtype C Env in a randomized controlled clinical trial. Vaccine. 2023 Apr 17;41(16):2696-2706. doi: 10.1016/j.vaccine.2023.03.015. Epub 2023 Mar 17. PMID 36935288